CLINICAL TRIAL: NCT04175977
Title: The Hospice Advanced Dementia Symptom Management and Quality of Life Trial (HAS-QOL) Stepped Wedge Trial
Brief Title: The Hospice Advanced Dementia Symptom Management and Quality of Life Trial (HAS-QOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-01186; 5R33AG061904-05 (NIH)
Record Dates: First submitted 2019-11-12; First posted 2019-11-25 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Wave 1: Usual Care for Months 1-7, Transition for Months 8-9, Intervention for Months 10-26 (Experimental): PWD at the hospice sites randomized to Wave 1 will receive usual care for 7 months, followed by the 2-month-long transition to the intervention over months 8 and 9, followed by the QAPI intervention for 16 Months from Month 10-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 2: Usual Care for Months 1-8, Transition for Months 9-10, Intervention for Months 11-26 (Experimental): PWD at the hospice sites randomized to Wave 2 will receive usual care for 8 months, followed by the 2-month-long transition to the intervention over months 9 and 10, followed by the QAPI intervention for 15 months from Month 11-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 3: Usual Care for Months 1-9, Transition for Months 10-11, Intervention for Months 12-26 (Experimental): PWD at the hospice sites randomized to Wave 3 will receive usual care for 9 months, followed by the 2-month-long transition to the intervention during months 10 and 11, followed by the QAPI intervention for 14 months from Months 12-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 4: Usual Care for Months 1-10, Transition for Months 11-12, Intervention for Months 13-26 (Experimental): PWD at the hospice sites randomized to Wave 4 will receive usual care for 10 months, followed by the 2-month-long transition to the intervention during months 11 and 12, followed by the QAPI intervention for 13 months from Months 13-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 5: Usual Care for Months 1-11, Transition for Months 12-13, Intervention for Months 14-26 (Experimental): PWD at the hospice sites randomized to Wave 5 will receive usual care for 11 months, followed by the 2-month-long transition to the intervention during months 12 and 13, followed by the QAPI intervention for 12 months from Months 14-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 6: Usual Care for Months 1-12, Transition for Months 13-14, Intervention for Months 15-26 (Experimental): PWD at the hospice sites randomized to Wave 6 will receive usual care for 12 months, followed by the 2-month-long transition to the intervention during months 13 and 14, followed by the QAPI intervention for 11 months from Months 15-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 7: Usual Care for Months 1-13, Transition for Months 14-15, Intervention for Months 16-26 (Experimental): PWD at the hospice sites randomized to Wave 7 will receive usual care for 13 months, followed by the 2-month-long transition to the intervention during months 14 and 15, followed by the QAPI intervention for 10 months from Months 16-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care
- Wave 8: Usual Care for Months 1-14, Transition for Months 15-16, Intervention for Months 17-26 (Experimental): PWD at the hospice sites randomized to Wave 7 will receive usual care for 14 months, followed by the 2-month-long transition to the intervention during months 15 and 16, followed by the QAPI intervention for 9 months from Months 17-26.
  Interventions: Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Aliviado Dementia Care-Hospice Edition QAPI program — Multi-modal QAPI program for improving the quality of care provided to PWD and support to their informal caregivers through hospice. It has been culturally tailored for use in diverse settings and tested with multiple minority communities in New York, including multiple Hispanic groups and African-Americans and Caribbean blacks. The intervention includes mentorship, training, a toolkit, and mobile app to assist clinicians in providing evidence-based symptom management to persons with dementia.
Behavioral: Usual Care — Usual care as provided by the hospice agency

SUMMARY:
The Aliviado Dementia Care Program (formerly known as the Dementia Symptom Management at Home Program, or DSM-H) was developed to implement dementia friendly care for persons with Dementia and their caregivers living in the community. Aliviado Dementia Care-Hospice Edition is a systems level quality assurance performance improvement program that includes interdisciplinary team training, validated assessment instruments, patient-centered care plans, treatment algorithms for behavioral and psychological symptoms of dementia and terminal delirium, and caregiver education pamphlets. Utilizing the R61/R33 mechanism, the Aliviado Dementia Care-Hospice Edition was successfully implemented in 2 sequential pilot trials in the hospice setting in 2019 (R61 phase). Following the successful pilot trials and the attainment of the R61 milestones, the investigators now seek to test the effectiveness of Aliviado Dementia Care-Hospice Edition in a pragmatic RCT in 25 hospice agencies across the nation (R33 phase) on its ability to reduce antipsychotic use (primary outcome) and effect quality (secondary and exploratory outcomes).

DETAILED DESCRIPTION:
As the population ages, the incidence rate of Alzheimer's Disease and Related Disorders (dementia) is expected to triple. The National Alzheimer's Plan recognizes that while the number of persons with dementia (PWD) is increasing substantially, the healthcare and long term care systems are unprepared to provide high quality, effective and efficient care to the PWD and their caregivers. PWD often have many behavioral and psychological symptoms of dementia (BPSD) including agitation, depression and sleep disturbances that affect both the quality of life (QOL) of the PWD and the caregiver. Unfortunately, due to a lack of programs to insert evidence-based care into the community, and hospice system specifically, PWD receive inappropriate and even harmful care. The investigators have developed the Aliviado Dementia Care Program (formerly known as the Dementia Symptom Management at Home Program, or DSM-H) to implement dementia friendly care for PWD and their caregivers in the community. Initially developed for use in home healthcare (HHC), the investigators have modified the program for use in hospice. The Aliviado Dementia Care-Hospice Edition is a systems level quality assurance performance improvement (QAPI) program that includes workforce training, and agency level workflow changes.

ELIGIBILITY:
Inclusion Criteria:

Interdisciplinary Team (IDT) MEMBERS:

* All English speaking IDT members
* Employed or contracted by the participating agency who are receiving Aliviado Dementia Care-Hospice Edition online or champion training
* All PWD (Persons with dementia) who are newly admitted to a participating hospice during the timeframe following implementation of the intervention who are over the age of 50 and have an ICD-10 code corresponding to a dementia diagnosis in their chart will be eligible.
* Greater than 18 years of age

Exclusion Criteria:

IDT MEMBERS:

• IDT members who are per diem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44143 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Monthly Percentage of Home Hospice Patients who are Prescribed Antipsychotic Medication | Baseline, Month 26
  Antipsychotic use measured using medical records.
Change from Baseline in Monthly Percentage of Home Hospice Patients who are Prescribed Non-Opioid Analgesic Medication | Baseline, Month 26
  Non-opioid analgesic use measured using medical records.

SECONDARY OUTCOMES:
Change from Baseline in Monthly Hours of Continuous Hospice Use | Baseline, Month 26
  Measured using hospice administrative data.
Change from Baseline in Monthly Days of Inpatient Hospice Use | Baseline, Month 26
  Measured using hospice administrative data.
Change from Baseline in Monthly Days of Respite Care | Baseline, Month 26
  Measured using hospice administrative data.
Change from Baseline in Monthly Percentage of Participants who are Permanently Institutionalized in a Nursing Home | Baseline, Month 26
  Measured using hospice administrative data.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Brody, Ph.D., Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).Upon reasonable request. Requests should be directed to Abraham.Brody@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Lin SY, Schneider CE, Bristol AA, Clancy M, Sprague SA, Aldridge M, Cortes T, Goldfeld KS, Kutner JS, Mitchell SL, Shega JW, Wu B, Zhu CW, Brody AA. Findings of Sequential Pilot Trials of Aliviado Dementia Care to Inform an Embedded Pragmatic Clinical Trial. Gerontologist. 2022 Feb 9;62(2):304-314. doi: 10.1093/geront/gnaa220. PMID 33377138